CLINICAL TRIAL: NCT04496193
Title: Comparing the Effects of Adding Dexamethasone in 0.25% Ropivacaine With 0.5% Ropivacaine Alone in the Quadratus Lumborum Block
Brief Title: The Effects of Adding Dexamethasone in the Quadratus Lumborum Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20200099
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-06

CONDITIONS: Analgesia; Motor Activity
MeSH Terms: conditions — Agnosia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group lower dose ropivacaine with dexamethasone (Experimental): Quadratus lumborum block was administered with 0.25% Ropivacaine 20 ml + dexamethasone 0.8 ml (4mg) at the end of surgery
  Interventions: Procedure: Quadratus Lumborum block
- Group higher dose ropivacaine with N/S (Active Comparator): Quadratus lumborum block was administered with 0.5% Ropivacaine 20 ml + N/S 0.8 ml at the end of surgery
  Interventions: Procedure: Quadratus Lumborum block
- Group lower dose ropivacaine with N/S (Placebo Comparator): Quadratus lumborum block was administered with 0.25% Ropivacaine 20 ml + N/S 0.8 ml at the end of surgery
  Interventions: Procedure: Quadratus Lumborum block

INTERVENTIONS:
Procedure: Quadratus Lumborum block — Quadratus Lumborum block is a type of plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle with the goal of anesthetizing the thoracolumbar nerves.

SUMMARY:
The quadratus lumborum block is widely used in abdominal surgery for post-operative analgesia. It is now also used for pain relief after hip surgery. Under the traditional blocking method, a high concentration of long-acting local anesthetic is used in order to achieve a long-term blocking effect. However, this is also likely to cause the patient's quadriceps weakness during the block period, increasing the risk of the patient falling during rehabilitation. It also increases systemic local anesthetic poisoning and may even trigger the risk of serious side effects such as cardiac arrest. Ropivacaine is a novel long-acting topical amine anesthetics that lasts long and has anesthetic and analgesic effects. Its pharmacological characteristics are low cardiotoxicity, sensory block and motor block separation at low concentrations more obvious, and with the external peripheral vasoconstriction. Therefore, the drug is especially suitable for postoperative analgesia.

Dexamethasone is a synthetic corticosteroid for the treatment of a wide range of symptoms including rheumatic diseases, certain skin diseases, severe allergies, asthma, chronic obstructive pulmonary disease, cerebral edema, and may also be combined with antibiotics for tuberculosis patients. It is becoming more common to use steroids as an adjuvant to local anesthetics in peripheral nerve block. Steroids have neurological blockade effects by blocking the nociceptive transmission of pith-type C-fibers and inhibiting the release of ectopic neurons. Dexamethasone, as a local anesthetic adjuvant in peripheral nerve block, has also been widely studied recently.

In order to reduce the incidence of long-acting topical anesthetics from the nerve block in the quadratus lumborum block, reducing the local anesthetic concentration is a feasible method. However, this will also result in a shorter time to neurological block. The investigators hypothesized that the addition of Dexamethasone 5 mg to low concentrations (0.25%) of Ropivacaine would prolong postoperative analgesia. Therefore, the purpose of this study was to compare the postoperative analgesia and the side effects of postoperative quadratus lumborum block with the addition of Dexamethasone 4mg to Ropivacaine (0.25%) in low concentrations and Ropivacaine (0.5%) alone.

DETAILED DESCRIPTION:
Test drug:

1. Name: Dexamethasone sod. Phosphate
2. Dosage form: 5 milligram (mg)/1 milliliter (mL)/Amp
3. Dose(s): 4mg
4. Dosing schedule: Dexamethasone 4mg adds into 0.25% Ropivacaine 20 mL
5. Mechanism of action: Synthesis of adrenocortical hormones, has a strong anti-inflammatory effect, can prolong the effect of local anesthetic drugs
6. Pharmacological category: HS051 Glucocorticoids

Study design:

1. ☑ Control: ☑ placebo（N/S 0.8 mL + 0.25% Ropivacaine 20 mL）

* active (Dexamethasone 4mg＋0.25% Ropivacaine 20 mL)
* others（N/S 0.8 mL + 0. 5% Ropivacaine 20 mL） □ Uncontrolled 2. Blinding: □ open-label □ single blind ☑ double blind □ others 3. Randomized: ☑ yes □ no 4. ☑ Parallel □ cross-over □ others 5. Duration of study：from Institutional Review Board (IRB) approval ~to 12, 31, 2022 ,total 24 months Duration of Enrollment : from IRB approval ~to 12, 31, 2022 ,total 24 months Duration of treatment：from IRB approval ~to 12, 31, 2022 ,total 24 months Duration of follow-up: from IRB approval ~to 12, 31, 2022 ,total 24 months

  * Multi-national □multi-center(Taiwan) ☑single center(Taiwan) 6. Number of subjects: 90 7. Is there any of the followings included Data Safety and Monitoring Board (DSMB)
  * yes ☑ no

Assessment criteria:

1. Efficacy:

1. The intensity of pain was assessed using a 0 to 10 Numerical Rating Scale (NRS) to quantify their degree of pain; where 0 means no pain and 10 the worst pain imaginable.
2. The analgesic activity was assessed using standard measures during the 48-hour treatment period: baseline pain intensity, time to rescue medication, and overall patient evaluation of study medication.

2. Safety:

1. Record the hemodynamic parameters during the 60-minute observation period in the anesthesia recovery room.
2. The severity of postoperative side effects (nausea, vomiting, pruritus) was quantified using different scales. Other side effects, including dizziness and drowsiness, are also recorded.
3. Motor block is assessed using Modified Bromage Scale.

3. Pharmacokinetics: None

4. Quality of life:

1. analgesic activity and duration of action
2. patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification: I ~ III
* Patients who received quadratus lumborum block for post-hip surgery analgesia

Exclusion Criteria:

* Lumbar plexus degeneration,
* Coagulation abnormalities with international normalized ratio (INR) > 1.5
* Obvious heart, lung, liver or kidney disease
* Body mass index less than 18.5 or greater than 35
* Pregnancy
* Regular use of steroids or opiates Opioids
* Chronic medication or alcohol abuse
* Previous allergies or adverse reactions to opiates, dexamethasone, or ropivacaine

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the post-operative analgesic effect of quadratus lumborum block | Within 48 hours after surgery
  1. The pain will be assessed using a 0 to 10 Numerical Rating Scale (NRS)
  2. In an hour in the recovery room, the pain will be evaluated every 15 minutes.
  3. Then the pain will be assessed at the 3rd, 6th, 12th, 24th, 36th, and 48th hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, MD, PhD, Principal Investigator — Department of Anesthesiology, Kaohsiung Medical University Hospital